CLINICAL TRIAL: NCT01037920
Title: An Intervention to Improve Communication Between Physicians and Minority Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: R21HL089623 (NIH)
Record Dates: First submitted 2009-12-18; First posted 2009-12-23 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): subjects in the intervention arm will complete a self-affirmation exercise prior to a physician visit
  Interventions: Behavioral: Self-affirmation exercise
- Control (Active Comparator): subjects in the intervention arm will complete a sham exercise prior to a physician visit
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Self-affirmation exercise — The intervention exercise asks subjects to reflect on a list of 11 personal values and to circle 2 or 3 items that are most important to them. Subjects are asked then to write a few sentences to describe why they are important.
  Arms: Intervention
Behavioral: Control — The control exercise is the same as the intervention exercise except that subjects reflect and write about values important to someone else.
  Arms: Control

SUMMARY:
The objective of the project is a test-of-concept of an intervention to reduce the effects of the perception of discrimination on the care of patients with chronic illness. Perception of discrimination manifests itself as stereotype threat. We hypothesize that stereotype threat impairs communication between minority patients and their physicians because of increased stress and diminished trust, resulting in interactions that are less successful at enhancing patient self-efficacy, in turn resulting in lower rates of adherence with anti-hypertensive medication.

The intervention is a self-affirmation exercise performed prior to a patient-physician visit. A similar intervention has been shown to reduce the racial gap in academic performance in middle school classrooms.

We will explore the mechanistic effects of the intervention by analysis of audiotapes of patient-provider visits following the intervention. We will measure the effect of the intervention on minority hypertensive patients' adherence with antihypertensive medication and blood pressure.

We will enroll 200 African American and Latino patients with hypertension and randomize 100 patients to perform the exercise and 100 patients to perform a null control exercise before the visit. We will assess change in patient's adherence with antihypertensive medications and in blood pressure over the six months following the index visit. In order to better understand the effects of the intervention we will measure subject's mood following the exercise, and self-reported stress levels, trust in the physician, and medication self-efficacy following the visit. We will also assess the quality of the patient-provider interaction from detailed analysis of audiotapes and from patient questionnaires. Following a subsequent patient-physician visit, we will conduct telephone interviews with patients to assess for persistence of any effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hypertension
* age > 21 years
* use of Denver Health as their usual source of care and pharmacy services
* self-described race/ethnicity of African American or Latino
* ability to provide informed consent

Exclusion Criteria:

* pregnancy-related hypertension
* end-stage renal disease
* unable to speak or write English at at least a 6th grade level.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
medication adherence | 6 months

SECONDARY OUTCOMES:
Blood pressure | 3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Derived] Havranek EP, Hanratty R, Tate C, Dickinson LM, Steiner JF, Cohen G, Blair IA. The effect of values affirmation on race-discordant patient-provider communication. Arch Intern Med. 2012 Nov 26;172(21):1662-7. doi: 10.1001/2013.jamainternmed.258. PMID 23128568